CLINICAL TRIAL: NCT02719626
Title: Improving The Safety And Nutritional Adequacy Of The Home Food Supply Of Elderly Recipients Of Home Delivered Meals
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 10-551Mx; USDA NIFSI # 2010-51110-21078 (Other Grant/Funding Number: USDA NIFSI)
Record Dates: First submitted 2016-02-03; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Food Safety; Nutritive Value; Homebound Persons; Frail Elderly
Keywords: senior; nutrition; home delivered meals; food safety; emergency prep

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Rutgers University will partner with the Meals on Wheels America (MOWA) and affiliated agencies in five states to conduct a study designed to improve food safety nutrition and emergency preparedness among homebound elderly recipients of home delivered meals (HDM). This population is at increased risk for food borne diseases, as a result of unique physiological and behavioral factors, and is particularly vulnerable to any disruptions in the food system because of their lack of mobility.

A multi-method research approach will be used with a target sample of 1,000 MOWA homebound elderly clients. Methods include the use of a novel UPC scanning technology that quickly and comprehensively catalogues all of the food in the clients' homes, a home food safety audit, and a face-to-face interview.

The goal of the study is to provide an improved understanding of the unique food safety threats to this at-risk population, suggest easy, cost-effective ways of reducing known food safety risk factors, and provide clear guidelines about the amount and types of food most needed by this population in emergency situations. Dissemination of research findings and recommendations will be done through a partnership with EDEN and MOWA, both of which have national constituencies poised to act on the recommendations.

DETAILED DESCRIPTION:
Elderly homebound recipients of home delivered meals (HDM) are at increased risk for foodborne disease and particularly vulnerable to disruptions that might prevent the delivery or safe consumption of food. In addition, there is a great deal of variability in the cognitive and physical abilities of those within this population, as well as a range of access to financial resources and social support that may vary both individually and geographically. Moreover, the agencies serving this population depend heavily on the time and donations of volunteers to carry out their important work. Therefore, to ensure their implementation, interventions designed to address food safety issues within this population must be relatively simple, efficient, and cost effective.

To address these issues, a multi-method research approach will be used, incorporating Universal Product Code (UPC) scanning technology combined with a dynamically growing database of foods and their associated nutritional parameters to catalogue the in-home food supply, an extant home food safety audit form, modified for study use, and a computer-enhanced questionnaire administered during an in-home interview. This project will provide a useful understanding of the nutritional and food safety gaps in this at-risk population that will allow for the design and testing of interventions to improve the food safety of both the HDM and the in-home food available to the homebound elderly. It will also provide clear and useful guidelines about the amount and types of food most needed by this population in emergency situations. Dissemination of the resulting research findings and recommendations will be accomplished through a partnership with the Extension Disaster Education Network (EDEN) and MOWA, both of whom have national constituencies poised to act on the recommendations.

HDM agencies from 5 states (AR, CA, IA, NJ, SC) will be purposively selected because of the varied characteristics of their HDM clients, as identified in an analysis of HDM recipients by state. The purposive sample of states included at least one from each of four of the quintiles on the MOWA Senior Hunger state ranking, with two states from the top quintile. The chosen states also represented a range in terms of the percentage minority clients, with some high in minority population and one extremely low. Finally, the percentage of rural clients ranged from zero in one state to almost 70% in another. Each of the five agencies will be asked to complete the study protocol with 200 eligible HDM recipients drawn from those on their client rolls using random numbers generated by the study investigators. Sampling with replacement will be carried out until a quota of 200 participants is reached, or no additional eligible clients can be recruited within each agency. A targeted sample size of 200 participants for each agency was selected to provide an overall target sample of 1000 HDM recipients to yield an overall sampling error rate of ± 3.1%, based on a population of approximately 900,000 HDM recipients.

The study:

1. Will analyze the food safety and quality parameters of the home food environments of homebound elderly recipients of HDM, and identify specific barriers to safe food-handling and storage practices by members of this high risk population. Refrigerator/freezer temperatures will be taken and adjustment made as needed to ensure that refrigerated foods are stored below 40 °F and frozen foods below 0 °F.
2. Will estimate the nutrient density and adequacy of the home food supplies of homebound elderly recipients of HDM, and identify areas of nutrition in which this population is deficient and would benefit from specific supplemental nutrition, especially during emergencies.
3. Two interventions will be proposed to improve food safety in homebound elderly recipients of HDM: the implementation of dating labels on the meals to help prevent the consumption of potentially unsafe older foods; checking refrigerator/freezer temperatures to determine temperature adherence/ maintenance, with adjustment made as needed.
4. Will partner with nutritionists, emergency preparedness experts, MOWA, and the Extension Disaster Education Network (EDEN) to develop and disseminate food safety and emergency preparedness recommendations specifically tailored to the needs of the homebound elderly. Materials will be developed for emergency food providers, home delivery meal providers and the elderly themselves.

Rutgers will partner with the Meals on Wheels America (MOWA) and selected MOWA affiliated agencies in five states to conduct an in-depth study of this vulnerable population designed to improve the nutrition and safety of food consumed by homebound elderly recipients of HDM, and to strengthen the nation's food defense system by identifying and addressing the critical nutrition needs of this population, particularly during times of emergency.

ELIGIBILITY:
Inclusion Criteria:

* 60 or more years old
* live alone
* no overt cognitive impairment
* receiving home delivered meals for at least 6 months prior to the in-home visit

Exclusion Criteria:

* < 60 years old
* do not live alone
* overt cognitive impairment
* receiving home delivered meals for less than 6 months prior to the in-home visit

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Home delivered meal recipients for at least 6 months, who: live alone, are 60 or more years old, have no overt cognitive impairment, and are from 5 states (AR, CA, IA, NJ & SC; one site per state).
Sampling Method: Non-Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Food Safety Kitchen Audit Score | Day 1
  A 7-scale home food safety kitchen audit score was calculated by summing the affirmative responses to the audit questions was calculated for each household. Items on each scale ranged from 3-12 for total score of 0 to 43 and all were weighted equally.
Nutritional Adequacy Ratio (NAR) | Day 1
  A household Nutrition Adequacy Ratio was calculated by summing nutrition values based on the daily values for a 2,000kcal diet for each food. NARs are ratios where 1 is recommended, >1 is more than recommended and <1 is inadequate.

SECONDARY OUTCOMES:
Nutritional Quality Score (QS) | Day 1
  A household summary nutrition quality score was calculated by summing up the NARs for 6 recommended nutrients and dividing the result by the NARs for the non-recommended nutrients in the home food supply for each household.
  Quality Score is a ratio where 1 is recommended, >1 is more than recommended and <1 is inadequate.

CONTACTS AND LOCATIONS:
Overall Officials: William K Hallman, PhD, Principal Investigator — Department of Human Ecology, Rutgers the State University of New Jersey; Carol Byrd-Bredbenner, PhD, RD, Principal Investigator — Department of Nutrition, Rutgers the State University of New Jersey
Locations (7):
- United States (7):
  - CareLink, Little Rock, Arkansas
  - St. Vincent's Meals on Wheels, Los Angeles, California
  - The Heritage Agency on Aging, Cedar Rapids, Iowa
  - Linden Meals on Wheels, Linden, New Jersey
  - Rutgers University, New Brunswick, New Jersey
  - Greenville Meals on Wheels, Greenville, South Carolina
  - Meals on Wheels America, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: No
Aggregate results will be made available via website (in process).

REFERENCES:
- [Background] Albertson AM, Wold AC, Joshi N. Ready-to-Eat Cereal Consumption Patterns: The Relationship to Nutrient Intake, Whole Grain Intake, and Body Mass Index in an Older American Population. J Aging Res. 2012;2012:631310. doi: 10.1155/2012/631310. Epub 2012 Oct 10. PMID 23094158
- [Background] Aldrich N, Benson WF. Disaster preparedness and the chronic disease needs of vulnerable older adults. Prev Chronic Dis. 2008 Jan;5(1):A27. Epub 2007 Dec 15. PMID 18082016
- [Background] Anderson AL, Verrill LA, Sahyoun NR. Food safety perceptions and practices of older adults. Public Health Rep. 2011 Mar-Apr;126(2):220-7. doi: 10.1177/003335491112600213. PMID 21387952
- [Background] Almanza BA, Namkung Y, Ismail JA, Nelson DC. Clients' safe food-handling knowledge and risk behavior in a home-delivered meal program. J Am Diet Assoc. 2007 May;107(5):816-21. doi: 10.1016/j.jada.2007.02.043. PMID 17467379
- [Background] Altshuler, N & Schimmel, J. USDHHS, Administration on Aging. Aging in Place: Do Older Americans Act Title III Services Reach Those Most Likely to Enter Nursing Homes? Research Brief Number 1, 2010. Available at: http://www.aoa.gov/aoaroot/program_results/docs/2010/AoA1_NursingHomes_012011.pdf Accessed on 06/23/14.
- [Background] Barile JP, Thompson WW, Zack MM, Krahn GL, Horner-Johnson W, Bowen SE. Multiple chronic medical conditions and health-related quality of life in older adults, 2004-2006. Prev Chronic Dis. 2013 Sep 26;10:E162. doi: 10.5888/pcd10.120282. PMID 24070034
- [Background] Barrett, A & Schimmel, J. USDHHS, Administration on Aging. OAA Title III Services Target the Most Vulnerable Elderly in the United States. Research Brief Number 2, 2010. Available at: http://www.aoa.gov/Program_Results/docs/2010/AoA_2_HealthStatus_041311.pdf Accessed on 06/23/2014.
- [Background] Blackburn ML, Bruhn CM, Miller LS, Ganthavorn C, Ober BA. Seniors, and their food handlers and caregivers, need food safety and nutrition education. Calif Agric. 2014;68(1):30-37. DOI: 10.3733/ca.v068n01p30.
- [Background] Bouillon K, Kivimaki M, Hamer M, Shipley MJ, Akbaraly TN, Tabak A, Singh-Manoux A, Batty GD. Diabetes risk factors, diabetes risk algorithms, and the prediction of future frailty: the Whitehall II prospective cohort study. J Am Med Dir Assoc. 2013 Nov;14(11):851.e1-6. doi: 10.1016/j.jamda.2013.08.016. Epub 2013 Oct 6. PMID 24103860
- [Background] Buzby JC. Older adults at risk of complications from microbial foodborne illness. Food Review. 2002;25(2):30-35.
- [Background] Byrd-Bredbenner C, Maurer J, Wheatley V, Cottone E, Clancy M. Food safety hazards lurk in the kitchens of young adults. J Food Prot. 2007 Apr;70(4):991-6. doi: 10.4315/0362-028x-70.4.991. PMID 17477272
- [Background] Byrd-Bredbenner C, Abbot JM, Cussler E. Nutrient profile of household food supplies of families with young children. J Am Diet Assoc. 2009 Dec;109(12):2057-62. doi: 10.1016/j.jada.2009.09.006. PMID 19942024
- [Background] Byrd-Bredbenner C, Schaffner DW, Maurer Abbot J. How food safe is your home kitchen? A self-directed home kitchen audit. J Nutr Educ Behav. 2010 Jul-Aug;42(4):286-9. doi: 10.1016/j.jneb.2010.01.008. No abstract available. PMID 20579613
- [Background] Cates SC, Kosa KM, Karns S, Godwin SL, Speller-Henderson L, Harrison R, Ann Draughon F. Food Safety Knowledge and Practices among Older Adults: Identifying Causes and Solutions for Risky Behaviors. J Nutr Elder. 2009 Apr;28(2):112-26. doi: 10.1080/01639360902949986. PMID 21184361
- [Background] Champion V & Skinner C. The Health Belief Model. In: Glanz K, Rimer B, Viswanath K, eds. Health behavior and health education: theory, research, and practice, 4th Ed. San Francisco: Jossey-Bass, 2008:45-66.
- [Background] Chobanian AV, Hill M. National Heart, Lung, and Blood Institute Workshop on Sodium and Blood Pressure : a critical review of current scientific evidence. Hypertension. 2000 Apr;35(4):858-63. doi: 10.1161/01.hyp.35.4.858. No abstract available. PMID 10775551
- [Background] Choi BC, Pak AW. A catalog of biases in questionnaires. Prev Chronic Dis. 2005 Jan;2(1):A13. Epub 2004 Dec 15. PMID 15670466
- [Background] Darmon P, Kaiser MJ, Bauer JM, Sieber CC, Pichard C. Restrictive diets in the elderly: never say never again? Clin Nutr. 2010 Apr;29(2):170-4. doi: 10.1016/j.clnu.2009.11.002. Epub 2009 Nov 22. PMID 19932533
- [Background] Dickinson A, Wills W, Meah A, Short F. Food safety and older people: the Kitchen Life study. Br J Community Nurs. 2014 May;19(5):226, 228-32. doi: 10.12968/bjcn.2014.19.5.226. PMID 24784557
- [Background] Donelson, SM; Murtaugh, CM; Feldman, PH; Hijjazi, K; Bruno, L; Zeppie, S; Neder, SK; Quint, E; Huang, L; Clark, A.. Clarifying the definition of homebound and medical necessity using OASIS data: Final report executive summary (2001). Center for Home Care Policy and Research. Available at: http://aspe.hhs.gov/daltcp/reports/2001/OASISfres.htm. Accessed on 03/21/2014.
- [Background] Drewnowski A, Fulgoni V 3rd. Nutrient profiling of foods: creating a nutrient-rich food index. Nutr Rev. 2008 Jan;66(1):23-39. doi: 10.1111/j.1753-4887.2007.00003.x. PMID 18254882
- [Background] Edfors E, Westergren A. Home-Living Elderly People's Views on Food and Meals. J Aging Res. 2012;2012:761291. doi: 10.1155/2012/761291. Epub 2012 Sep 9. PMID 22991667
- [Background] Evans EW, Redmond EC. Analysis of older adults' domestic kitchen storage practices in the United Kingdom: identification of risk factors associated with listeriosis. J Food Prot. 2015 Apr;78(4):738-45. doi: 10.4315/0362-028X.JFP-14-527. PMID 25836399
- [Background] Field A. Discovering Statistics Using IBM SPSS Statistics, 4th Edition SAGE Publications Ltd. Thousand Oaks, CA; 4th edition (January 24, 2013). IISBN-13: 978-1446249185.
- [Background] Fey-Yensan N, English C, Ash S, Wallace C, Museler H. Food safety risk identified in a population of elderly home-delivered meal participants. J Am Diet Assoc. 2001 Sep;101(9):1055-7. doi: 10.1016/S0002-8223(01)00259-0. No abstract available. PMID 11573760
- [Background] Fogler-Levitt E, Lau D, Csima A, Krondl M, Coleman P. Utilization of home-delivered meals by recipients 75 years of age or older. J Am Diet Assoc. 1995 May;95(5):552-7. doi: 10.1016/S0002-8223(95)00150-6. PMID 7722189
- [Background] Frewer L, Shepherd R, Sparks P. The interrelationship between perceived knowledge, control, and risk associated with a range of food-related hazards targeted at the individual, other people, and society. J Food Safety. 1994;14(1):19-40. DOI:10.1111/j.1745-4565.1994.tb00581.x
- [Background] Gerhard T. Bias: considerations for research practice. Am J Health Syst Pharm. 2008 Nov 15;65(22):2159-68. doi: 10.2146/ajhp070369. PMID 18997149
- [Background] GfK Social Research. Public Attitudes to Food Issues - Further analysis on those aged 65 and over. London: Food Safety Standards; 2009. Available at: http://tna.europarchive.org/20111116080332/http://www.food.gov.uk/multimedia/pdfs/pafiover65.pdf Accessed on 10/06/2015.
- [Background] Gollub EA, Weddle DO. Improvements in nutritional intake and quality of life among frail homebound older adults receiving home-delivered breakfast and lunch. J Am Diet Assoc. 2004 Aug;104(8):1227-35. doi: 10.1016/j.jada.2004.05.204. PMID 15281039
- [Background] Gopinath B, Flood VM, McMahon CM, Burlutsky G, Brand-Miller J, Mitchell P. Dietary glycemic load is a predictor of age-related hearing loss in older adults. J Nutr. 2010 Dec;140(12):2207-12. doi: 10.3945/jn.110.128462. Epub 2010 Oct 6. PMID 20926604
- [Background] Green AK, Jacques PF, Rogers G, Fox CS, Meigs JB, McKeown NM. Sugar-sweetened beverages and prevalence of the metabolically abnormal phenotype in the Framingham Heart Study. Obesity (Silver Spring). 2014 May;22(5):E157-63. doi: 10.1002/oby.20724. Epub 2014 Mar 8. PMID 24550031
- [Background] Guthrie HA, Scheer JC. Validity of a dietary score for assessing nutrient adequacy. J Am Diet Assoc. 1981 Mar;78(3):240-5. PMID 7217578
- [Background] He, W; Sengupta, M; Velkoff, VA; DeBarros, KA. 65+ in the United States: Washington (DC): U.S. Department of Health and Human Services, National Institutes of Health, National Institute on Aging, and U.S. Department of Commerce, Economics and Statistics Administration, U.S. Census Bureau; 2005. Available at: http://www.census.gov/prod/2006pubs/p23-209.pdf. Accessed on 04/22/14.
- [Background] Heron M. Deaths: leading causes for 2010. Natl Vital Stat Rep. 2013 Dec 20;62(6):1-96. PMID 24364902
- [Background] Kleinman R & Foster L. USDHHS, Administration on Aging. Multiple Chronic Conditions Among OAA Title III Program Participants. Research Brief Number 4, 2011. Available at: http://www.aoa.gov/aoaroot/program_results/docs/2011/AoA4_Chronic_508.pdf Accessed on 06/23/2014.
- [Background] Kosa KM, Cates SC, Godwin SL, Ball M, Harrison RE. Effectiveness of educational interventions to improve food safety practices among older adults. J Nutr Gerontol Geriatr. 2011;30(4):369-83. doi: 10.1080/21551197.2011.623943. PMID 22098179
- [Background] Kosa KM, Cates SC, Karns S, Godwin SL, Chambers D. Consumer home refrigeration practices: results of a web-based survey. J Food Prot. 2007 Jul;70(7):1640-9. doi: 10.4315/0362-028x-70.7.1640. PMID 17685337
- [Background] McGuire S. Institute of Medicine. 2010. Strategies to Reduce Sodium Intake in the United States. Washington, DC: The National Academies Press. Adv Nutr. 2010 Nov;1(1):49-50. doi: 10.3945/an.110.1002. Epub 2010 Nov 16. No abstract available. PMID 22043452
- [Background] Iuliano S, Olden A, Woods J. Meeting the nutritional needs of elderly residents in aged-care: are we doing enough? J Nutr Health Aging. 2013;17(6):503-8. doi: 10.1007/s12603-013-0042-7. PMID 23732545
- [Background] Jacobson MF, Havas S, McCarter R. Changes in sodium levels in processed and restaurant foods, 2005 to 2011. JAMA Intern Med. 2013 Jul 22;173(14):1285-91. doi: 10.1001/jamainternmed.2013.6154. PMID 23699927
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Franceschi S, Hamidi M, Marchie A, Jenkins AL, Axelsen M. Glycemic index: overview of implications in health and disease. Am J Clin Nutr. 2002 Jul;76(1):266S-73S. doi: 10.1093/ajcn/76/1.266S. PMID 12081850
- [Background] Johnson AE, Donkin AJ, Morgan K, Lilley JM, Neale RJ, Page RM, Silburn R. Food safety knowledge and practice among elderly people living at home. J Epidemiol Community Health. 1998 Nov;52(11):745-8. doi: 10.1136/jech.52.11.745. PMID 10396508
- [Background] Johnson DB, Beaudoin S, Smith LT, Beresford SA, LoGerfo JP. Increasing fruit and vegetable intake in homebound elders: the Seattle Senior Farmers' Market Nutrition Pilot Program. Prev Chronic Dis. 2004 Jan;1(1):A03. Epub 2003 Dec 15. PMID 15634365
- [Background] Joung HW, Kim HS, Yuan JJ, Huffman L. Service quality, satisfaction, and behavioral intention in home delivered meals program. Nutr Res Pract. 2011 Apr;5(2):163-8. doi: 10.4162/nrp.2011.5.2.163. Epub 2011 Apr 25. PMID 21556231
- [Background] Kamp BJ, Wellman NS, Russell C; American Dietetic Association; American Society for Nutrition; Society for Nutrition Education. Position of the American Dietetic Association, American Society for Nutrition, and Society for Nutrition Education: Food and nutrition programs for community-residing older adults. J Am Diet Assoc. 2010 Mar;110(3):463-72. doi: 10.1016/j.jada.2009.12.009. PMID 20213956
- [Background] Keller HH. Meal programs improve nutritional risk: a longitudinal analysis of community-living seniors. J Am Diet Assoc. 2006 Jul;106(7):1042-8. doi: 10.1016/j.jada.2006.04.023. PMID 16815120
- [Background] Kretser AJ, Voss T, Kerr WW, Cavadini C, Friedmann J. Effects of two models of nutritional intervention on homebound older adults at nutritional risk. J Am Diet Assoc. 2003 Mar;103(3):329-36. doi: 10.1053/jada.2003.50052. PMID 12616254
- [Background] Lund BM, O'Brien SJ. The occurrence and prevention of foodborne disease in vulnerable people. Foodborne Pathog Dis. 2011 Sep;8(9):961-73. doi: 10.1089/fpd.2011.0860. Epub 2011 May 11. PMID 21561383
- [Background] Martin-Biggers J, Yorkin M, Aljallad C, Ciecierski C, Akhabue I, McKinley J, Hernandez K, Yablonsky C, Jackson R, Quick V, Byrd-Bredbenner C. What foods are US supermarkets promoting? A content analysis of supermarket sales circulars. Appetite. 2013 Mar;62:160-5. doi: 10.1016/j.appet.2012.12.001. Epub 2012 Dec 8. PMID 23228904
- [Background] Millen BE, Ohls JC, Ponza M, McCool AC. The elderly nutrition program: an effective national framework for preventive nutrition interventions. J Am Diet Assoc. 2002 Feb;102(2):234-40. doi: 10.1016/s0002-8223(02)90055-6. PMID 11846117
- [Background] Morley JE. Decreased food intake with aging. J Gerontol A Biol Sci Med Sci. 2001 Oct;56 Spec No 2:81-8. doi: 10.1093/gerona/56.suppl_2.81. PMID 11730241
- [Background] MOW. History of Meals on Wheels Programs (2014).. Available at: http://www.nwsds.org/content/Senior%20Meals/History%20of%20Meals%20on%20Wheels%20Program.pdf Accessed on 11/19/2015.
- [Background] Nieuwenhuizen WF, Weenen H, Rigby P, Hetherington MM. Older adults and patients in need of nutritional support: review of current treatment options and factors influencing nutritional intake. Clin Nutr. 2010 Apr;29(2):160-9. doi: 10.1016/j.clnu.2009.09.003. Epub 2009 Oct 13. PMID 19828215
- [Background] NLEA. Nutrition Labeling and Education Act (1990). Available at, http://www.fda.gov/Food/GuidanceRegulation/GuidanceDocumentsRegulatoryInformation/LabelingNutrition/ucm2006828.htm Accessed on 03/21/14.
- [Background] NSF International. The Public Health and Safety Organization. Food expiration dates survey. Available at: http://www.nsf.org/consumer-resources/studies-articles/surveys/food-expiration-datessurvey Accessed on 09/16/2015.
- [Background] Older Americans. Federal Interagency Forum on Aging-Related Statistics. Older Americans 2012: Key Indicators of Well-Being. Federal Interagency Forum on Aging-Related Statistics. Washington, DC: U.S. Government Printing Office. June 2012. Available at: http://www.agingstats.gov/Main_Site/Data/2012_Documents/docs/EntireChartbook.pdf Accessed on 03/21/2014.
- [Background] Ouellette J & Wood W. Habit and intention in everyday life: the multiple processes by which past behavior predicts future behavior. Psychol Bulletin. 1998;124:54-74. DOI: 0033-2909198.
- [Background] Pouillot R, Hoelzer K, Jackson KA, Henao OL, Silk BJ. Relative risk of listeriosis in Foodborne Diseases Active Surveillance Network (FoodNet) sites according to age, pregnancy, and ethnicity. Clin Infect Dis. 2012 Jun;54 Suppl 5:S405-10. doi: 10.1093/cid/cis269. PMID 22572661
- [Background] Qiu WQ, Dean M, Liu T, George L, Gann M, Cohen J, Bruce ML. Physical and mental health of homebound older adults: an overlooked population. J Am Geriatr Soc. 2010 Dec;58(12):2423-8. doi: 10.1111/j.1532-5415.2010.03161.x. Epub 2010 Nov 10. PMID 21070195
- [Background] Quinlan JJ. Foodborne illness incidence rates and food safety risks for populations of low socioeconomic status and minority race/ethnicity: a review of the literature. Int J Environ Res Public Health. 2013 Aug 15;10(8):3634-52. doi: 10.3390/ijerph10083634. PMID 23955239
- [Background] Woodburn MJ, Raab CA. Household Food Preparers' Food-Safety Knowledge and Practices Following Widely Publicized Outbreaks of Foodborne Illness. J Food Prot. 1997 Sep;60(9):1105-1109. doi: 10.4315/0362-028X-60.9.1105. PMID 31207831
- [Background] Raab CA & Woodburn MJ. Changing risk perceptions and food-handling practices of Oregon household food preparers. Int J Consum Stud. & Home Economics. 1997;21(2): 117-130. DOI: 10.1111/j.1470-6431.1997.tb00274.x.
- [Background] Remond D, Shahar DR, Gille D, Pinto P, Kachal J, Peyron MA, Dos Santos CN, Walther B, Bordoni A, Dupont D, Tomas-Cobos L, Vergeres G. Understanding the gastrointestinal tract of the elderly to develop dietary solutions that prevent malnutrition. Oncotarget. 2015 Jun 10;6(16):13858-98. doi: 10.18632/oncotarget.4030. PMID 26091351
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):188-97. doi: 10.1161/CIR.0b013e3182456d46. No abstract available. PMID 22215894
- [Background] Rolls BJ. Do chemosensory changes influence food intake in the elderly? Physiol Behav. 1999 Apr;66(2):193-7. doi: 10.1016/s0031-9384(98)00264-9. PMID 10336143
- [Background] Roseman MG. Food safety perceptions and behaviors of participants in congregate-meal and home-delivered-meal programs. J Environ Health. 2007 Sep;70(2):13-21, 44. PMID 17886577
- [Background] Roseman MG & Hayek K. Determining the success of food safety education to elderly participating in congregate and home-delivered meal programs. J Am Diet Assoc. 2005;105(8), Supp.13. DOI: http://dx.doi.org/10.1016/j.jada.2005.05.029.
- [Background] Schefske SD, Bellows AC, Byrd-Bredbenner C, Cuite CL, Rapport H, Vivar T, Hallman WK. Nutrient analysis of varying socioeconomic status home food environments in New Jersey. Appetite. 2010 Apr;54(2):384-9. doi: 10.1016/j.appet.2010.01.007. Epub 2010 Jan 15. PMID 20079787
- [Background] Scheidt DM, Daniel E. Composite index for aggregating nutrient density using food labels: ratio of recommended to restricted food components. J Nutr Educ Behav. 2004 Jan-Feb;36(1):35-9. doi: 10.1016/s1499-4046(06)60126-7. PMID 14756980
- [Background] Schiffman SS. Effects of aging on the human taste system. Ann N Y Acad Sci. 2009 Jul;1170:725-9. doi: 10.1111/j.1749-6632.2009.03924.x. PMID 19686219
- [Background] Sharkey JR, Branch LG, Zohoori N, Giuliani C, Busby-Whitehead J, Haines PS. Inadequate nutrient intakes among homebound elderly and their correlation with individual characteristics and health-related factors. Am J Clin Nutr. 2002 Dec;76(6):1435-45. doi: 10.1093/ajcn/76.6.1435. PMID 12450914
- [Background] Smith JL. Foodborne illness in the elderly. J Food Prot. 1998 Sep;61(9):1229-39. doi: 10.4315/0362-028x-61.9.1229. PMID 9766083
- [Background] Stevens J, Bryant M, Wang L, Borja J, Bentley ME. Exhaustive measurement of food items in the home using a universal product code scanner. Public Health Nutr. 2011 Feb;14(2):314-8. doi: 10.1017/S1368980010001837. Epub 2010 Jul 6. PMID 20602866
- [Background] Tasevska N, Park Y, Jiao L, Hollenbeck A, Subar AF, Potischman N. Sugars and risk of mortality in the NIH-AARP Diet and Health Study. Am J Clin Nutr. 2014 May;99(5):1077-88. doi: 10.3945/ajcn.113.069369. Epub 2014 Feb 19. PMID 24552754
- [Background] Thermostatic Mixing Valve Manufacturers Association (TMVA). Recommended code of practice for safe water temperatures for infants and elderly. London: 2000. Available at: www.beama.org.uk/asset/022A6360-7B36-4F5B-A192238D9C4F896E/ Accessed on 03/03/2015.
- [Background] Thomas KS, Mor V. Providing more home-delivered meals is one way to keep older adults with low care needs out of nursing homes. Health Aff (Millwood). 2013 Oct;32(10):1796-802. doi: 10.1377/hlthaff.2013.0390. PMID 24101071
- [Background] Thomas KS, Mor V. The relationship between older Americans Act Title III state expenditures and prevalence of low-care nursing home residents. Health Serv Res. 2013 Jun;48(3):1215-26. doi: 10.1111/1475-6773.12015. Epub 2012 Dec 3. PMID 23205536
- [Background] Thomas KS & Dosa D. More Than a Meal: results from a March, 2015 pilot - a randomized control trial of home-delivered meal programs. Available at: http://www.mealsonwheelsamerica.org/theissue/facts-resources/more-than-a-meal Accessed on 09/13/2015.
- [Background] U.S. Census Bureau. National Population Projections: Table 3. Percent distribution of the projected population by selected age groups and sex for the United States: 2010 to 2050. Released 8/2008 (based on Census 2000). Washington, DC: U.S. Census Bureau. Available at: http://www.census.gov/population/projections/data/national/2008/summarytables.html Accessed on 03/21/2014.
- [Background] U.S. Census Bureau. DeNavas-Walt, C; Proctor, BD; Smith, JC. Current Population Reports, P60-239, Income, Poverty, and Health Insurance Coverage in the United States: 2010, U.S. Government Printing Office, Washington, DC. Available at: https://www.census.gov/prod/2011pubs/p60-239.pdf Accessed on 03/21/2014.
- [Background] U.S. Census Bureau. Annual estimates of the resident population by sex and selected age groups for the United States: July 1 2010 - 2012. Washington, DC: U.S. Census Bureau. Available at: https://www.census.gov/popest/data/national/asrh/2012/index.html; Accessed on 03/21/2014.
- [Background] U.S. Census Bureau. State & County: QuickFacts 2014. Available at: http://quickfacts.census.gov/qfd/states/00000.html Accessed on 09/19/2015.
- [Background] USDHHS, AoA. U.S Department of Health and Human Services, Administration on Aging: First national survey of older Americans act Title III service recipients 2002-2003. Available at: https://aoasurvey.org/docs/1st_highlights.pdf Accessed on 10/02/2015.
- [Background] USDHHS, AoA. U.S Department of Health and Human Services, Administration on Aging. Nutrition Services: Title IIIC2 Older Americans Act & Section 336. Available at: http://www.aoa.gov/AoA_programs/HCLTC/Nutrition_Services/index.aspx Accessed on 03/21/2014.
- [Background] USDHHS, AoA. U.S Department of Health and Human Services, Administration on Aging: Elderly nutrition program (2013). Available at: http://www.acl.gov/NewsRoom/Publications/docs/Elderly_Nutrition_Programs_1.pdf Accessed on 10/15/2015.
- [Background] USDHHS, ACL. U.S. Department of Health and Human Services, Administration for Community Living, Administration on Aging: Aging statistics. (2007). Available at: http://www.aoa.acl.gov/Aging_Statistics/Profile/2007/8.aspx Accessed on 09/19/2015.
- [Background] USDHHS, ACL. U.S Department of Health and Human Services, Administration for Community Living, Administration on Aging: Aging Statistics. (2014). Available at: www.aoa.acl.gov/Aging_Statistics/index.aspx Accessed on 09/19/ 2015.
- [Background] USDHHS, CDC. U.S Department of Health and Human Services, Centers for Disease Control and Prevention. A Cup of Health with CDC: More to Consider Than the Salt Shaker Sodium Intake: Quantities and Food Sources - United States, 2005-2006. Recorded: June 22, 2010; posted: July 1, 2010 Available at: http://www2c.cdc.gov/podcasts/media/pdf/mmwr5_070110_transcript.pdf Accessed on 05/08/2014.
- [Background] Centers for Disease Control and Prevention (CDC). Incidence and trends of infection with pathogens transmitted commonly through food - foodborne diseases active surveillance network, 10 U.S. sites, 1996-2012. MMWR Morb Mortal Wkly Rep. 2013 Apr 19;62(15):283-7. PMID 23594684
- [Background] USDHHS, CDC. U.S Department of Health and Human Services, Centers for Disease Control and Prevention. 2011 Estimates of foodborne illness in the United States. Available at: http://www.cdc.gov/foodborneburden/2011-foodborne-estimates.html Accessed on 09/15/2015.
- [Background] USDHHS, CDC. U.S. Department of Health and Human Services, Centers for Disease Control and Prevention. Healthy people 2020. Available at: http://www.healthypeople.gov/2020/topics-objectives/topic/food-safety Accessed on 12/05/2015.
- [Background] USDHHS, CMMS. U.S Department of Health and Human Services, Centers for Medicare & Medicaid Services. Medicare Benefit Policy Manual Chapter 7 - Home Health Services Rev. 208, 05-11-15 30.1.1 - Patient confined to the home (2015). Available at: https://www.cms.gov/Regulations-and-Guidance/Guidance/Manuals/Internet-Only-Manuals-Ioms-Items/Cms012673.html Accessed on 10/09/2015.
- [Background] USDHHS, FDA. U.S Department of Health and Human Services, U.S. Food and Drug Administration, Guide to nutrition labeling and education act (NLEA) requirements. Nutritional Labeling and Education Act (NLEA) Requirements (8/94 - 2/95). Office of Regulatory Affairs, U.S. Food & Drug Administration(1995). Available at: http://www.fda.gov/ICECI/Inspections/InspectionGuides/ucm074948.htm Accessed on 03/21/2014.
- [Background] USDHHS, FDA. U.S Department of Health and Human Services, U.S. Food and Drug Administration, Appendix F: Calculate the Percent Daily Value for the Appropriate Nutrients Guidance for Industry: A Food Labeling Guide - Guidance, Compliance & Regulatory Information (2008). Available at: http://www.fda.gov/Food/GuidanceComplianceRegulatoryInformation/GuidanceDocuments/FoodLabelingNutrition/FoodLabelingGuide/ucm064928.htm . Accessed on 03/21/2014
- [Background] USDHHS, FDA. U.S Department of Health and Human Services, U.S. Food and Drug Administration, Refrigerator thermometers: cold facts about food safety. Available at: http://www.fda.gov/food/foodborneillnesscontaminants/buystoreservesafefood/ucm253954.htm Accessed on 03/17/2015.
- [Background] USDHHS, FDA. U.S Department of Health and Human Services, U.S. Food and Drug Administration. Food safety: it's especially important for at-risk groups. Available at: http://www.fda.gov/Food/FoodborneIllnessContaminants/PeopleAtRisk/ucm352830.htm Accessed on 09/13/2015.
- [Background] USDHHS, FDA & USDA. U.S Department of Health and Human Services, U.S. Food and Drug Administration & U.S. Department of Agriculture - Food Safety and Inspection Service. Food Safety for people with diabetes: a need-to know guide for those who have been diagnosed with diabetes. 2011, Rev. Available at: http://www.fda.gov/Food/FoodborneIllnessContaminants/PeopleAtRisk/ucm312706.htm Accessed 11/02/2015.
- [Background] USDHHS, FDA & USDA. U.S Department of Health and Human Services, U.S. Food and Drug Administration & U.S. Department of Agriculture, Food safety for older adults. A need-to-know guide for those 65 years of age and older. Washington, DC: National Academy Press, 2011.
- [Background] USDHHS, USDA. U.S Department of Health and Human Services, U.S. Department of Agriculture ARS. Dietary guidelines for Americans, 7th Ed. Washington, DC: National Academy Press, 2010. Available at: http://www.cnpp.usda.gov/dgas2010-dgacreport.htm Accessed on 05/01/2014.
- [Background] USDHHS, IFSAC. U.S Department of Health and Human Services, Interagency Food Safety Analytics Collaboration (IFSAC) Project Report: Foodborne illness source attribution estimates for Salmonella, Escherichia coli O157 (E. coli O157), Listeria monocytogenes (Lm), and Campylobacter using outbreak surveillance data, February 2015. Available at: http://www.cdc.gov/foodsafety/pdfs/ifsac-project-report-508c.pdf Accessed on 09/15/2015.
- [Background] Vasan RS, Beiser A, Seshadri S, Larson MG, Kannel WB, D'Agostino RB, Levy D. Residual lifetime risk for developing hypertension in middle-aged women and men: The Framingham Heart Study. JAMA. 2002 Feb 27;287(8):1003-10. doi: 10.1001/jama.287.8.1003. PMID 11866648
- [Background] Weaver CM, Dwyer J, Fulgoni VL 3rd, King JC, Leveille GA, MacDonald RS, Ordovas J, Schnakenberg D. Processed foods: contributions to nutrition. Am J Clin Nutr. 2014 Jun;99(6):1525-42. doi: 10.3945/ajcn.114.089284. Epub 2014 Apr 23. PMID 24760975
- [Background] Weinstein JL, Phillips V, MacLeod E, Arsenault M, Ferris AM. A universal product code scanner is a feasible method of measuring household food inventory and food use patterns in low-income families. J Am Diet Assoc. 2006 Mar;106(3):443-5. doi: 10.1016/j.jada.2005.12.004. PMID 16503237
- [Background] Whelton PK, Appel LJ, Sacco RL, Anderson CA, Antman EM, Campbell N, Dunbar SB, Frohlich ED, Hall JE, Jessup M, Labarthe DR, MacGregor GA, Sacks FM, Stamler J, Vafiadis DK, Van Horn LV. Sodium, blood pressure, and cardiovascular disease: further evidence supporting the American Heart Association sodium reduction recommendations. Circulation. 2012 Dec 11;126(24):2880-9. doi: 10.1161/CIR.0b013e318279acbf. Epub 2012 Nov 2. PMID 23124030
- [Background] WHO. World Health Organization/Food and Agricultural Organization of the United Nations. Diet, nutrition, and the prevention of chronic diseases. Available at: http://www.who.int/dietphysicalactivity/publications/trs916/download/en/index.html. Accessed on 03/21/2014.
- [Background] WHO. World Health Organization Forum on Reducing Salt Intake in Populations. (2008). Reducing Salt Intake in Populations: Report of a WHO Forum and Technical Meeting 5-7 October 2006, Paris, France. Geneva, Switzerland: World Health Organization; 2008. Available at: http://www.who.int/dietphysicalactivity/Salt_Report_VC_april07.pdf Accessed on 04/22/2014.
- [Background] Ziliak JP, Gundersen C. Senior hunger in the United States: differences across states and rural and urban areas. A report submitted to Meals On Wheels Association of America, Inc. September 2009. Internet: http://www.nfesh.org/research/ Accessed on 11/02/2015.